CLINICAL TRIAL: NCT00189176
Title: Phase I/II Trial of Tetrathiomolybdate (TM) in Patients With Usual Interstitial Pneumonia Refractory to Previous Therapy
Brief Title: Safety Study of Tetrathiomolybdate in Patients With Idiopathic Pulmonary Fibrosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Coalition for Pulmonary Fibrosis (Unknown)
Responsible Party: Principal Investigator, Kevin R. Flaherty, Associate Professor of Medicine, University of Michigan
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2002-0806
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-02

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — tetrathiomolybdate

ARMS (1):
- Tetrathiomolybdate (Experimental)
  Interventions: Drug: Tetrathiomolybdate

INTERVENTIONS:
Drug: Tetrathiomolybdate

SUMMARY:
This study will evaluate the safety of the administration of a copper chelating agent, tetrathiomolybdate, for patients with idiopathic pulmonary fibrosis that have failed previous treatment. The primary endpoint for this study is safety with secondary endpoints including change in pulmonary function, exercise capacity, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic pulmonary fibrosis
* Disease progression despite six months of treatment (steroids with/without azathioprine or cyclophosphamide) defined by at least one of the following:

  * Increased symptoms
  * Decline in forced vital capacity of at least 10%
  * Decline in diffusion capacity for carbon monoxide of at least 20%
  * Increased infiltrate on CXR or high resolution CT scan
* Taking < 15 mg prednisone for at least 30 days prior to screening
* Age 35-80, inclusive
* Able to understand a written informed consent and comply with the study protocol

Exclusion Criteria:

* Significant environmental exposure
* Diagnosis of collagen vascular disease
* Evidence of active infection
* Clinically significant cardiac disease:

  * Myocardial infarction, coronary artery bypass or angioplasty within 6mo
  * Unstable angina pectoris
  * Congestive heart failure requiring hospitalization within 6 months
  * Uncontrolled arrhythmia
* Poorly controlled or severe diabetes mellitus
* Pregnancy or lactation
* Women of childbearing potential not using a medically approved means of contraception (i.e. oral contraceptives, intrauterine devices, diaphragm, Norplant)
* Current enrollment in another experimental protocol

Physiologic Criteria:

* FEV1/FVC < 0.60

Laboratory Criteria:

* Total bilirubin > 1.5 X upper limit normal
* AST or ALT > 3X upper limit normal
* Alkaline phosphatase > 3X upper limit normal
* White blood cell count < 2,500/mm3
* Hematocrit < 30%
* Platelets < 100,000/mm3
* Prothrombin time INR > 1.5

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2003-03; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Safety | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kevin R Flaherty, MD, MS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States